CLINICAL TRIAL: NCT03974568
Title: Evaluation of Peripheral Perfusion Index as a Predictor of Failure of Weaning From Mechanical Ventilation
Brief Title: Peripheral Perfusion Index in Weaning From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, assistant professor, Cairo University
Other Study IDs: N-159-2018
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — arterial blood gases (ABG)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral perfusion index (PPI) is variable measured by Radical-7 (Masimo) device and reflects the ratio between pulsatile and non-pulsatile portions of peripheral circulation. PPI is characterized by being non-invasive, real time, and simple variable. Impairment of various perfusion indices (such as central venous oxygen saturation and serum lactate) during spontaneous breathing trial (SBT) were previously reported; however, these indices are characterized by being relatively invasive. We hypothesized that impairment of PPI during SBT might be predictive of weaning failure. The aim of this work was to evaluate the possible association between PPI and success of SBT

DETAILED DESCRIPTION:
This prospective observational study will be carried out in surgical intensive care unit (SICU) unit of trauma and emergency hospital at Cairo University teaching hospital. Informed consent will be obtained from patients' next-of-kin prior to the enrolment in the study. All mechanically ventilated patients for more than 48 hours presented will be consecutively included.

The excluded patients are: patients < 18 years, patients with peripheral vascular disease, patients on vasopressors, and those with hand injuries hindering which would preclude the application of the device probe will be excluded.

Assessment of readiness to wean from mechanical ventilation will be done by ICU physician according to the ICU protocol Spontaneous breathing trial (SBT) will be applied through pressure support (PS) mode with PS 5 cmH2O and positive end expiratory pressure (PEEP) 5 cmH2O for 30 minutes; then, weaning parameters will be assessed again. The decision of extubation will be taken by the intensivist in charge who is blinded to peripheral perfusion index (PPI) measurements. Weaning failure will be defined according to the guidelines of international conference on weaning from mechanical ventilation PPI will be continuously monitored using Radical-7 device pulse co-oximeter (Masimo corporation, Irvine, CA) via a pulse oximeter probe applied to the third or fourth digit of left hand. The probe will be covered with an opaque shield to avoid any error by external light sources. A baseline reading for PPI will be obtained followed by a reading each 5 minutes till the end of the SBT. We calculated a PPI ratio to evaluate the change in PPI during SBT. PPI ratio is defined as PPI by the end of SBT / baseline PPI).

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients for more than 48 hours

Exclusion Criteria:

* patients < 18 years
* patients with peripheral vascular disease
* patients on vasopressors
* patients with hand injuries hindering which would preclude the application of the device probe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
peripheral perfusion index (PPI) ratio | 30 minutes
  PPI by the end of spontaneous breathing trial (SBT) / baseline PPI

SECONDARY OUTCOMES:
peripheral perfusion index | 30 minutes
  ratio between pulsatile and non-pulsatile portions of peripheral circulation
heart rate | 30 minutes
  beat per minutes
systolic blood pressure | 30 minutes
  mmHg
cardiac output | 30 minutes
  litre/minutes
central venous pressure | 30 minutes
  cmH2O
respiratory rate | 30 minutes
  breath per minutes
Rapid shallow breathing index | At end of 30 minutes of SBT
  respiratory rate / tidal volume

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lotfy A, Hasanin A, Rashad M, Mostafa M, Saad D, Mahmoud M, Hamimy W, Fouad AZ. Peripheral perfusion index as a predictor of failed weaning from mechanical ventilation. J Clin Monit Comput. 2021 Apr;35(2):405-412. doi: 10.1007/s10877-020-00483-1. Epub 2020 Feb 8. PMID 32036499